CLINICAL TRIAL: NCT00592254
Title: A Screening Protocol for Adults With Attention Deficit Hyperactivity Disorder
Brief Title: Screening Protocol for Adults With ADHD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Other Study IDs: 2002-P-001856
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: ADHD
Keywords: ADHD; Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A

SUMMARY:
The objective of this protocol is to establish a comprehensive screening process to evaluate the eligibility of potential adult subjects for appropriate ADHD clinical research studies

DETAILED DESCRIPTION:
To address the needs of the large number of adults who contact the Adult ADHD Program at Massachusetts General Hospital annually, we have sought approval for several research studies aimed at evaluating critical components of the needs of this population. Potential participants for those studies present with a widely varied set of complaints not always discernable in a telephone screening interview. This state of affairs often makes it difficult to ask subjects to sign a specific protocol's consent form without obtaining additional clinical information. Because of this, we have potential subjects consent to undergo an in-depth clinical assessment that will allow them to be screened by a clinician for eligibility to a diverse clinical research program available to them.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18-55
2. Subjects must have a DSM-IV or DSM-V diagnosis of ADHD, as determined by a clinical evaluation based on DSM-IV or DSM-V criteria

Exclusion Criteria:

1. History of head trauma with loss of consciousness, organic brain disorders, seizures, or neurosurgical intervention.
2. Any significant medical condition, in the judgment of the investigator
3. Mental retardation
4. Pregnancy of lactation
5. Subjects with a known recent history (within the past 6 months) of illicit drug or alcohol dependence
6. Sensory difficulties such as deafness or blindness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with symptoms of ADHD
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2002-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Screening Protocol | Sreening
  This study is a prescreening for possible entry into other studies

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html